CLINICAL TRIAL: NCT04768426
Title: Phase II Trial of Circulating Tumor DNA Monitoring During Adjuvant Capecitabine in Patients With Triple-negative Breast Cancer and Residual Disease Following Standard Neoadjuvant Chemotherapy
Brief Title: Serial Circulating Tumor DNA (ctDNA) Monitoring During Adjuvant Capecitabine in Early Triple-negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-57723; NCI-2021-01757 (Other: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2021-02-19; First posted 2021-02-24 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Triple Negative Breast Cancer; Breast Cancer
Keywords: TNBC; Triple Negative Breast Cancer; Post neoadjuvant; Residual disease; Capecitabine
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Neoplasm, Residual | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Capecitabine (Experimental): 1000 mg/m2 administered on Days 1 to 14 of 21-day cycles
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — 1000 mg/m2 administered on Days 1 to 14 of 21-day treatment cycles, for 8 cycles.
  Other Names: fluoropyrimidine carbamate

SUMMARY:
The purpose of the study is to evaluate the use of a circulating tumor DNA (ctDNA) assay, ie, a "liquid biopsy," as a tool to identify triple-negative breast cancer (TNBC) patients who will or will not experience benefit from treatment with capecitabine. Participants will be monitored for changes in ctDNA in the blood over time received during capecitabine treatment. Results of ctDNA analysis will be correlated to genetic characteristics of individual tumors. This may inform future clinical trials in which patients could receive a different treatment than capecitabine to reduce their risk of breast cancer relapse.

DETAILED DESCRIPTION:
The Primary Objective is to characterize the circulating tumor DNA (ctDNA) profile of triple-negative breast cancer (TNBC) in participants with residual disease after standard neoadjuvant chemotherapy (NAC) receiving standard-of-care adjuvant capecitabine.

The Secondary Objectives are to correlate ctDNA levels with genomic features and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Anatomic stage I - III triple-negative breast cancer at diagnosis
2. Estrogen receptors (ER) and Progesterone receptors (PR) status <10%
3. Residual disease following at least 4 cycles of neoadjuvant chemotherapy. Patients who received other investigational immunotherapy or targeted therapy during the neoadjuvant phase of treatment are eligible.
4. ≥ 18 years of age
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
6. All clinically significant toxic effects of prior cancer therapy resolved to Grade ≤ 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE, v 5.0), except alopecia and G2 neuropathy.
7. No evidence of metastatic disease.
8. A minimum 4-week wash out from previous chemotherapy treatment is required.
9. Adequate hematologic function: Absolute neutrophil count (ANC) ≥ 1,500 cells/μL (≥ 1,500/mm3); Platelets ≥ 100,000 cells/μL (≥ 100,000/mm3)
10. Adequate hepatic function: Bilirubin ≤ 1.5 times the specific institutional upper limit of normal (ULN). Exception: If Gilbert's syndrome; then ≤ 5 times ULN. Aspartate transaminase (AST) and alanine transaminase (ALT) each ≤ 2.5 x ULN
11. Adequate renal function: Serum creatinine ≤ 1.5 x ULN; or calculated creatinine clearance > 50 mL/min using the Cockcroft Gault formula.
12. Planned for 6 months or 8 cycles of adjuvant capecitabine.
13. Women of childbearing potential (WOCBP) must have a negative pregnancy test.
14. WOCBP must agree to use effective contraception during the study and for 3 months after the last dose.
15. Male participants and their female partners of child bearing potential must be willing to use an appropriate method of contraception during the study and for 3 months after the last dose.
16. Capable of giving signed informed consent, which includes compliance with requirements and restrictions listed in the informed consent form (ICF) and in the protocol

Exclusion Criteria:

1. Metastatic breast cancer
2. Has not had definitive surgical resection
3. Pregnant or breastfeeding
4. Has not completed definitive adjuvant radiation if planned
5. Known human immunodeficiency virus (HIV) positivity or active hepatitis B or C.
6. Investigational agents within 4 weeks of study initiation
7. Inability to swallow oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Baseline levels of ctDNA detection | 6 months
  In participants with triple-negative breast cancer (TNBC) who have received standard neoadjuvant chemotherapy (NAC), levels of circulating tumor DNA (ctDNA) will be assessed at baseline and after 6 months of standard adjuvant capecitabine treatment. The outcome will be reported as the number of participants who are:
  * ctDNA+ (ctDNA-positive) at baseline and at 6 months.
  * ctDNA+ at baseline but ctDNA- (ctDNA-negative) at 6 months.
  * ctDNA- at baseline and at 6 months.
  * ctDNA- at baseline but ctDNA+ at 6 months.
  The outcome is a number without dispersion.

SECONDARY OUTCOMES:
Correlation of ctDNA levels with genomic features of tumor | 24 weeks
  Genomic status of certain mutations in the tumor will be assessed by next-generation sequencing in participants who are:
  * ctDNA+ (ctDNA-positive) at baseline and at 6 months.
  * ctDNA+ at baseline but ctDNA- (ctDNA-negative) at 6 months.
  * ctDNA- at baseline and at 6 months.
  * ctDNA- at baseline but ctDNA+ at 6 months.
  The genes of interest are:
  PIK3CA AKT AKT1 PTEN BRCA1 BRCA2 PALB2 CHEK2 ATM NBN BRIP1 BARD1 MRE11 ATR RAD50 RAD51C RAD51D FANCA FANCC FANCD2 FANCE FANCF FANCG FANCL.
  The outcome will be reported as the number of participants with a positive mutation status in the gene of interest. The outcome is a number without dispersion.
Overall Survival (OS) | 5 years
  Overall survival (OS) will be assessed as participants remaining alive 5 years from the first treatment initiation. The outcome is reported as the number of participants alive (without dispersion).
Relapse-Free Survival | 5 years
  Relapse-free survival is defined as the time from treatment initiation to first invasive relapse or death, through 5 years. The outcome is reported as the number of participants with relapse-free survival (without dispersion) at 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Telli, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No